CLINICAL TRIAL: NCT01291485
Title: Randomized Clinical Trial Examining the Efficacy of an Electronic Intervention for HIV Medication Adherence
Brief Title: Electronic Intervention for HIV Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Kasey Claborn, Doctoral Candidate, Oklahoma State University Center for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2010022
Record Dates: First submitted 2011-01-10; First posted 2011-02-08 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: HIV
Keywords: HIV; Medication adherence; computer-based intervention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): Intervention includes education about HIV and medication adherence, motivational interviewing, cognitive behavioral techniques, and problem-solving strategies to improve HIV medication adherence and clinical outcomes.
  Interventions: Behavioral: Life Steps for Medication Adherence
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Life Steps for Medication Adherence — The intervention was adapted into an electronic version of the empirically supported Life Steps intervention for HIV medication adherence. Education about HIV and medication adherence, motivational interviewing, cognitive behavioral techniques, and problem-solving strategies to improve medication adherence and clinical outcomes in people living with HIV were also included in the intervention.
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to develop and examine the feasibility and initial efficacy of a computer-based intervention to improve medication adherence among people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* infected with HIV
* over age 18
* currently prescribed a Highly Active Antiretroviral Therapy (HAART) regimen
* prescribed a regimen for the first time, changing regimens, or report adherence below 95% agree to brief follow-up interviews

Exclusion Criteria:

* physical impairment that would prevent them from successfully completing the computer-based program (e.g., blind, deaf, severe neuropsychological impairment)
* Actively psychotic
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HIV medication adherence | up to 6 months
  Self-reported adherence to HIV medications will be assessed using the AACTG Medication Adherence Questionnaire (M. A. Chesney, et al., 2000).

SECONDARY OUTCOMES:
HIV Treatment Adherence Self-Efficacy | Baseline, 1-month, 3 months, and 6-months
  Self-efficacy for adherence to HIV medications will be assessed using the HIV-ASES (Johnson et al., 2007). The HIV-ASES is a 12-item scale of patient confidence in their ability to carry out behaviors related to adhering to medication regimens. Responses range from 1 ("cannot do it at all") to 10 ("completely certain can do it"). Item scores are averaged with higher scores indicating higher adherence self-efficacy.
Quality of Life | Baseline, 1-month, 3-months, and 6-months
  Quality of life will be assessed using the McGill Quality of Life questionnaire (S. Robin Cohen, Hassan, Lapointe, & Mount, 1996). This instrument is a 16-item scale that assesses quality of life in four domains: physical well-being, psychological well-being, existential well-being, and support; each item is assessed on a 0-10 point scale.
Viral Load | Baseline, 1 month, 3 months, and 6 months
CD4 cell count | Baseline, 1 month, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thad R Leffingwell, Ph.D., Study Director — Oklahoma State University; Kasey R Claborn, M.S., Principal Investigator — Oklahoma State University; Johnny Stephens, Pharm.D., Study Chair — Oklahoma State University Center for Health Sciences
Locations (1):
- Internal Medicine Specialty Services, Tulsa, Oklahoma, United States